CLINICAL TRIAL: NCT03520699
Title: Beijing Friendship Hospital Metabolic Surgery Clinical Database
Brief Title: Beijing Friendship Hospital Metabolic Surgery Database
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigator, Beijing Friendship Hospital
Other Study IDs: BFH-MSD
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Surgery
Keywords: metabolic surgery; metabolic disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic surgery, as a recognition treatment option for patients with clinical morbid obesity, is gaining increasing appreciation. In addition to substantial weight loss, emerging studies have highlighted that metabolic surgery can substantially ameliorate obesity-related metabolic diseases, including but not limited to type 2 diabetes mellitus (T2DM), hypertension, dyslipidemia, obstructive sleep apnea-hypopnea syndrome (OSAHS) and polycystic ovary syndrome (PCOS)in severely obese patients. However, further investigations with larger sample size and longer observation time still needed to clarity the efficacy and safety of metabolic surgery in Chinese patients with obesity and encouraging future research in this field.

ELIGIBILITY:
Inclusion Criteria:

* be able to receive metabolic surgery (LSG or LRYGB)

Exclusion Criteria:

* can not be able to understand and willing to participate in this registry with signature

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with morbid obesity who are suitable and willing to accept metabolic surgical procedure and also agree with the registry
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the excess weight loss effect of metabolic surgery after 1year | 1 year after surgery
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)

SECONDARY OUTCOMES:
the adverse events rate of metabolic surgery | 30 days after surgery
  show the surgical safety by 30 days follow-up according to guideline（such as: bleeding, leak, obstruction, re-operation for complication）
the excess weight loss effect of metabolic surgery with long-time follow-ups | 3 years
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)
the excess weight loss effect of metabolic surgery with long-time follow-ups | 5 years
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)
the excess weight loss effect of metabolic surgery with long-time follow-ups | 10 years
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)
the glycemic control effect of metabolic surgery with long-time follow-ups | 3 years
  the decrease of HbA1c, glucose level, C-peptide and insulin levels
the glycemic control effect of metabolic surgery with long-time follow-ups | 5 years
  the decrease of HbA1c, glucose level, C-peptide and insulin levels
the glycemic control effect of metabolic surgery with long-time follow-ups | 10 years
  the decrease of HbA1c, glucose level, C-peptide and insulin levels
the glycemic control effect of metabolic surgery after 1 year | 1 year after surgery
  the decrease of HbA1c, glucose level, C-peptide and insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, China

REFERENCES:
- [Derived] Lv H, Li M, Liu Y, Zhao L, Sun J, Cao D, Zeng N, Liu J, Liu Y, Bian S, Zhang P, Yang Z, Zhang Z, Wang Z. The Clinical Value and Appropriateness Criteria of Upper Abdominal Magnetic Resonance Examinations in Patients Before and After Bariatric Surgery: a Study of 837 Images. Obes Surg. 2020 Oct;30(10):3784-3791. doi: 10.1007/s11695-020-04688-w. PMID 32483745
- [Derived] Zhang P, Liu Y, Lv H, Li MY, Yu FX, Wang Z, Ding HY, Wang LX, Zhao KX, Zhang ZY, Zhao PF, Li J, Yang ZH, Zhang ZT, Wang ZC. Integration of Neural Reward Processing and Appetite-Related Signaling in Obese Females: Evidence From Resting-State fMRI. J Magn Reson Imaging. 2019 Aug;50(2):541-551. doi: 10.1002/jmri.26576. Epub 2019 Jan 17. PMID 30653786